CLINICAL TRIAL: NCT04508218
Title: Impact of Adding Protein Supplementation to Exercise Training on Lean Body Mass and Muscle Strength in Burn Patients
Brief Title: Protein Supplementation and Exercise Training in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nesma Morgan Allam, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002758
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Burns
Keywords: Exercise training; Protein supplementation; Muscle strength; Lean body mass; Burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Protein+ Exercise group (Experimental): Received oral protein supplementation, exercise program and traditional burn care
  Interventions: Dietary Supplement: whey protein supplementation powder (Inkospor X-TREME; France); Other: Exercise training program; Other: traditional burn care
- Protein group (Experimental): Received oral protein supplementation and traditional burn care
  Interventions: Dietary Supplement: whey protein supplementation powder (Inkospor X-TREME; France); Other: traditional burn care
- Exercise group (Experimental): Received exercise program and traditional burn care
  Interventions: Other: Exercise training program; Other: traditional burn care
- Control group (Other): Received traditional burn care
  Interventions: Other: traditional burn care

INTERVENTIONS:
Dietary Supplement: whey protein supplementation powder (Inkospor X-TREME; France) — Protein requirements for burned adults are estimated as 1.5-2.0 g/kg/day. The participants asked to take the calculated serving of whey protein dissolved in 150ml of water two times / day in the morning and in the evening
  Arms: Protein group; Protein+ Exercise group
Other: Exercise training program — After healing of the burn (6 weeks after injury), participants in group A and group C started resisted exercise program with a qualified therapist for 1 hour three times/week on nonconsecutive days over 12 weeks. In addition, aerobic exercises were conducted on the treadmill. Peak oxygen consumption was assessed for all patients by using the exercise test on treadmill before participation in aerobic exercises.
  Arms: Exercise group; Protein+ Exercise group
Other: traditional burn care — ROM exercises, stretching, ADL activities and scar management

SUMMARY:
Burn injury causes continuous catabolism of the skeletal muscle resulting in decreased muscle strength, muscle mass and impairment of functional mobility. Purpose: The purpose of this study is to investigate the efficacy of combination of exercise training and protein supplementation on lean body mass (LBM) and muscle strength in patients with severe burn.

DETAILED DESCRIPTION:
Sixty participants with severe burn > 30% total body surface area (TBSA) were randomly distributed into 4 equal groups of 15 participants per group. Group A (Protein+ Exercise group) received oral protein supplementation, exercise program and traditional burn care, group B (Protein group) received oral protein supplementation and traditional burn care, group C (Exercise group) received exercise program and traditional burn care, group D (Control group) received traditional burn care. LBM was measured using Dual-energy x-ray absorptiometry (DXA) while muscle strength was measured using Biodex 3 Dynamometer System before treatment and 12 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* healed deep partial-thickness thermal burn
* > 30% of TBSA and
* the exercise program started after healing of the burn (after burn injury by 6 weeks)

Exclusion Criteria:

* conditions that may affect on participation in the exercise program as a recent coronary disease, uncontrolled hypertension, orthopedic problems limiting exercise, abnormal cardiac stress test, pregnant women, refusal to participate in a physical activity program,
* presence of psychological or cognitive disorders (aggressive behavior, impulsivity, dementia)
* food intolerance to milk protein products.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
lean body mass | after 12 week of intervention
  The QDR 4500A densitometry system DXA (Hologic Inc., Bedford, USA) was used according to the manufacturer instructions for calculating LBM

SECONDARY OUTCOMES:
muscle strength | after 12 week of intervention
  The Biodex 3 Dynamometer Medical System (Shirley, USA) was utilized for strength assessment of quadriceps muscle of the dominant leg (concentric test) of the participants. It was performed according to manufacturer instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Nesma M Allam, PhD, Principal Investigator — lecturer at faculty of physical therapy
Locations (1):
- Nesma Morgan Allam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
results of the study
Supporting Information: Study Protocol
Time Frame: 6 months after puplication
Access Criteria: study protocol